CLINICAL TRIAL: NCT01515774
Title: An Open-label, Randomized, Multi-center, Crossover Study to Observe the Effect of Once-daily Mirapex ER® and Twice-daily Mirapex ER® in Patients With Parkinson Disease
Brief Title: Study to Observe the Effect of Mirapex ER® Once-daily (QD) Versus Twice-daily (BID)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-1104-062-358
Record Dates: First submitted 2012-01-10; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Pramipexole
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Give QD dose first then BID dosing
  Interventions: Drug: Mirapex ER
- Group 2 (Active Comparator): Give BID dosing and then QD dosing
  Interventions: Drug: Mirapex ER

INTERVENTIONS:
Drug: Mirapex ER — Change Requip or Mirapex to Mirapex ER

SUMMARY:
1. In order to observe the benefit, side effects, and patient preference of Mirapex ER when used in once-daily (QD) or twice-daily (BID) dosing
2. In order to estimate the conversion rate of dopamine agonists into Mirapex ER

DETAILED DESCRIPTION:
1. Study subjects : Parkinson disease who are on Requip or Mirapex and are considering to change into Mirapex ER
2. Cross over study design:

   * Group 1: Once daily dose for 2 month then into BID in divided dose for 2 months
   * Group 2: BID in divided dose for 2 months then into QD dose for 2 months
3. Dose adjustment may be done in the first 4 weeks.
4. Compare the benefit, side effects, and patient preference between the QD vs BID dosing

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30-80
2. Parkinson disease
3. On dopamine agonists (Requip or Mirapex) and are considering to change into Mirapex ER
4. On stable antiparkinsonian medication for at least 4 weeks
5. Who signed consent to the study

Exclusion Criteria:

1. Who are on less than 2 mg of Requip or 0.375 mg of Mirapex
2. Who have dementia, psychosis, major depression and other serious neurological or medical problems
3. Who are allergic to the similar medications
4. Who has history of heavy metal poisoning
5. Who were on othe clinical trials of other medications within the last 4 weeks
6. Who are pregnant or lactating
7. Who are considered not eligible by the investigator

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-08 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Patient preference | 4 months
  Overall preference in QD versus BID

SECONDARY OUTCOMES:
Motor complications | 2 months at each arm
  Visual rating scale for off severity, dyskinesia severity Duration - off duration, dyskinesia duration
Sleep problems | 2 months at each arm
  Parkinson's disease sleep scale (PDSS) Excessive daytime sleepiness scale(ESS)
Motor UPDRS and HY stage | 2months at each arm
Side effects | 2 months at each arm
  Rating scale (0~10): Nausea, Dizziness, Somnolence, Headache, Constipation, Dyspepsia, Fatigue, Hallucination, Edema, Dry mouth,Others
Patient global impression for improvement | 2 months at each arm
Preference in each factor | 4 months
  Preference of QD versus BID in each factor: off duration, off severity, dyskinesia duration, dyskinesia severity, on quality, adverse events, sleep quality, convenience
Patient choice | 4 months
  Patient choice in QD or BID Reason for the choice

CONTACTS AND LOCATIONS:
Overall Officials: Beom S Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Jenner P, Konen-Bergmann M, Schepers C, Haertter S. Pharmacokinetics of a once-daily extended-release formulation of pramipexole in healthy male volunteers: three studies. Clin Ther. 2009 Nov;31(11):2698-711. doi: 10.1016/j.clinthera.2009.10.018. PMID 20110012
- [Background] Rascol O, Barone P, Hauser RA, Mizuno Y, Poewe W, Schapira AH, Salin L, Sohr M, Debieuvre C; Pramipexole Switch Study Group. Efficacy, safety, and tolerability of overnight switching from immediate- to once daily extended-release pramipexole in early Parkinson's disease. Mov Disord. 2010 Oct 30;25(14):2326-32. doi: 10.1002/mds.23262. PMID 20669265
- [Derived] Yun JY, Kim YE, Yang HJ, Kim HJ, Jeon B. Twice-Daily versus Once-Daily Pramipexole Extended Release Dosage Regimens in Parkinson's Disease. Parkinsons Dis. 2017;2017:8518929. doi: 10.1155/2017/8518929. Epub 2017 Feb 7. PMID 28265478